CLINICAL TRIAL: NCT05839158
Title: Evaluation of the Efficacy of Follicles-derived Microtissue Homogenate in Promoting Wound Healing After Hair Transplantation
Brief Title: Evaluation of the Effect of HFMT in Promoting Donor-site Wound Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NFEC-2022-500
Record Dates: First submitted 2023-04-10; First posted 2023-05-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Wound Heal
Keywords: hair transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFMT treated (Experimental): The experimental group will receive treatment with HFMT ointment prepared in a homogenized mixture, applied once immediately after surgery to the treatment area.
  Interventions: Other: HFMT cell suspension
- Mupirocin treated (Placebo Comparator): The control group will receive treatment with Mupirocin applied once immediately after surgery to the control area.
  Interventions: Other: Mupirocin ointment

INTERVENTIONS:
Other: HFMT cell suspension — Perform FUE autologous hair transplantation on the patient according to the guidelines and standard procedures. During the procedure, a hollow punch is used to individually punch out follicular units from the donor area. The epidermis, some dermis tissue, sebaceous glands, and surrounding tissue of the follicular units are separated and removed before the remaining follicular tissue is implanted into the recipient area. The separated tissue is trimmed with surgical scissors to create a cell suspension. After completion of the procedure, the HFMT cell suspension is evenly applied to the treatment group surface. Double vaseline gauze is used to cover all donor areas and is then wrapped with sterile dry gauze with moderate pressure.
  Arms: HFMT treated
Other: Mupirocin ointment — the Minoxidil ointment is evenly applied to the control group surface.
  Arms: Mupirocin treated

SUMMARY:
Autologous hair transplantation involves follicle extraction, trimming, and implantation. Follicle trimming improves efficiency and postoperative appearance, resulting in the discarded tissue known as hair follicle-derived microtissue (HFMT). In a clinical case, HFMT homogenate was applied to the FUE donor area wound, resulting in reduced pain, relief from itching, and faster healing compared to conventional treatment. This study aims to compare the effects of HFMT on FUE donor area wound healing.

DETAILED DESCRIPTION:
The process of autologous hair transplantation involves three steps: FUE follicle extraction, follicle trimming, and follicle implantation. The purpose of follicle trimming is to improve the efficiency of follicle implantation and enhance the immediate postoperative aesthetic appearance. Therefore, during the follicle trimming process, the sebaceous glands and above-mentioned epidermis, partial dermis tissue, and surrounding tissue of the follicles are usually separated and discarded, and the remaining follicle tissue is implanted into the recipient area. The investigator collectively refers to the discarded tissue as hair follicle-derived microtissue (HFMT). In a clinical case, The investigator accidentally discovered that if the HFMT obtained from the follicular unit extraction (FUE) method was collected, cut into pieces, and made into tissue homogenate, and then the HFMT homogenate was used to cover the FUE donor area wound, the patient reported reduced postoperative pain and some relief from skin itching. Additionally, compared to conventionally treated wounds, the wound in the donor area healed faster. Based on these findings, this study aims to compare the effects of HFMT on the healing of FUE donor area wounds.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-60 years who underwent FUE autologous hair transplantation.
* The patient's liver and kidney function were normal, and the serum protein level before surgery was normal.

Exclusion Criteria:

* Patients with a history of smoking.
* Those suffering from diseases that affect wound healing, such as diabetes or hyperglycemia.
* Those with abnormal blood sugar.
* Abnormal cardiopulmonary function.
* There are foci of infection in or near the surgical area.
* Scar hyperplasia or scar constitution.
* Those with a history of neuralgia.
* The patient took immunosuppressants, cytostatics, and hormonal anticoagulants before surgery and antibiotics.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in the area of the wound at the donor site | post op days 3, 5, 7, 14 and post op weeks 4, 6, 8, 12, 16, 24
  Using a dermatoscope, randomly select 3 fields of view, measure the area of all wounds in the field of view, and calculate the average value of the deviation between the wound area and the initial wound area.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiqi Hu, MD, PhD, Study Chair — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The age of the participants and photographs of the skin under the dermatoscope will be presented in the paper
Supporting Information: Study Protocol, SAP, CSR
Time Frame: These data will continue to be presented in the paper after its publication.
Access Criteria: People with access to journal databases can access the relevant data of this study.